CLINICAL TRIAL: NCT03202433
Title: Use of Virtual Reality in Blood Donors, an Innovative Tool
Brief Title: Reduce Stress Associated With Needle Aspiration, in Voluntary and Replacement Blood Donors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Blood and Tissues IV and V Region, Chile (Other)
Responsible Party: Principal Investigator, Adrián Erich Goecke Varela, Medical Technologist, Center for Blood and Tissues IV and V Region, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORD1083
Record Dates: First submitted 2017-06-18; First posted 2017-06-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Stress
Keywords: Virtual Reality; Stress Reduction; Needle Aspiration; Blood Donors; Intervention

STUDY DESIGN:
Intervention Model Description: Allocation of two groups (Study and Control)
Who Masked: Outcomes Assessor
Masking Description: Blocks swapped.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Distractor (Experimental): The objective is to apply a technique, using virtual reality lenses, with relaxing audio-visual contents of no more than ten minutes, to reduce stress before and during the blood donation process and to respond to the level of pain perceived during donation, either post-puncture and withdrawal of the needle
  Interventions: Device: Use of virtual reality lenses, with relaxing audio-visual contents
- Traditional Blood Donation Process (No Intervention): The objective is to respond to the level of pain perceived during donation, either post-puncture and withdrawal of the needle, without virtual reality support

INTERVENTIONS:
Device: Use of virtual reality lenses, with relaxing audio-visual contents — Use of virtual reality lenses (and audio) as a distraction for the blood donor patients.
  Arms: Virtual Reality Distractor

SUMMARY:
Reduce stress associated with needle aspiration, in voluntary and replacement blood donors.

This study has not been completed.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effectiveness of Virtual Reality (as a form of distraction) to reduce the stress associated with extraction needle puncture in the volunteer blood donors and reposition of Fixed Collection of the Valparaiso Blood Center, Of the Valparaíso San Antonio Health Service.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and / or visualize the numerical scale of pain
* Spanish spoken
* Greater than 50 Kilograms of weight
* Blood hemoglobin: Greater than 12.5 g% in women and greater than 13.5 g% in men
* Have been accepted as a blood donor.

Exclusion Criteria:

* Unable to understand and / or visualize the numerical scale of pain
* Does not speak Spanish
* Less than 50 Kilograms
* Blood hemoglobin: Less than 12.5 g% in women and less than 13.5 g% in men.
* Have been rejected as a blood donor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-12-30; Primary Completion 2017-11-24 (Actual); Study Completion 2017-11-24

PRIMARY OUTCOMES:
Numerical scale of pain (EN) | Once finalized the donation that should last a maximum of 15 minutes.
  Main measure for pain perception

SECONDARY OUTCOMES:
Heart rate. Measurement with automatic equipment | Before donating, after the puncture and after the extraction of the needle.Maximum duration of the procedure, 15 minutes
  Measure for the perception of stress
Blood pressure. Measurement with automatic equipment | Before donating, after the puncture and after the extraction of the needle.Maximum duration of the procedure, 15 minutes
  Measure for the perception of stress

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Meneses, Study Director — Medical College of Chile
Locations (1):
- Blood and Tissue Center, Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riva G, Raspelli S, Pallavicini F, Grassi A, Algeri D, Wiederhold BK, Gaggioli A. Interreality in the management of psychological stress: a clinical scenario. Stud Health Technol Inform. 2010;154:20-5. PMID 20543263
- [Background] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- Available data/document: Clinical Study Report — http://www.researchgate.net/publication/287542931_Psychological_coping_with_invasive_and_painful_medical_procedures_in_the_treatment_of_childhood_and_adolescent_cancer_The_cognitive-behavioural_approach
- Available data/document: Study Protocol: ISSN 0124-8146 — http://scielo.org.co/scielo.php?script=sci_arttext&pid=S0124-81462013000200010
- Available data/document: Clinical Practice Guide — http://www.criscancer.org